CLINICAL TRIAL: NCT06079619
Title: Comparison of Dermatoscopy X400 Interpreted by 6 Non-dermatologists (3 Gynecologists, 3 General Practitioners) and an Artificial Intelligence Software Skin Artificial Intelligence Versus Dermatoscopy x 20 Interpreted by 3 Expert Dermatologists, for the Identification of 150 Genital Pigmented Tumors: Towards a New Medical Organization of the Dermatologist, Non-dermatologist Articulation?
Brief Title: Comparison of Dermatoscopy X400 Interpreted by 6 Non-dermatologists and an Artificial Intelligence Software Skin Artificial Intelligence Versus Dermatoscopy x 20
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN252022/CHUSTE
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2023-09

CONDITIONS: Genital Tumor; Pigmented Lesions
Keywords: dermoscopy; non-invasive imaging; melanotic macule; melanoses; mucosa; melanoma; vulva; glans; tumor; genital tumor; nevus
MeSH Terms: conditions — Melanosis; Melanoma; Neoplasms; Nevus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: expert dermatologists: Group A is composed of expert dermatologists. Group A doctors will have at their disposal 150 dermoscopic photos, x20 dermatoscopic photos according to the usual practice of pigmented genital tumors.
  The dermatologists will characterize the dermatoscopy with a standardized reading grid to assess the different dermatoscopic patterns of genital tumors.
  Interventions: Other: Analysis of photos of pigmented tumours by the three groups
- Group B: non-dermatologists: Group B is composed of gynecologists (Group B1) and general practitioners (B2) Group B physicians will only perform dermatoscopy x 400. They will have been given a maximum of 1 hour's training to identify melanosis-type pigmented tumors, which are the most frequent benign tumors in x 400 dermatoscopy.
  Only three x400 dermatoscopy patterns will be presented to them to the exclusion of all others, which are sufficient to identify benign lesions.
  Interventions: Other: Analysis of photos of pigmented tumours by the three groups
- Group C: Artificial intelligence: Artificial intelligence: the skin Artificial intelligence software, a learning base will be provided, different from the evaluation base and the test base.
  Interventions: Other: Analysis of photos of pigmented tumours by the three groups

INTERVENTIONS:
Other: Analysis of photos of pigmented tumours by the three groups — Analysis of photos of pigmented tumours by the three groups with different techniques for each group to compare them.

SUMMARY:
Pigmented lesions of the genital mucosa are common, affecting between 10% and 20% of the population. The clinical appearance is sometimes confusing. They are often extensive, irregular, and inhomogeneous in color, which can make them look suspicious. Moreover, dermatoscopic imaging is often complex to interpret, as shown by the many different patterns reported in the literature.

Thus, preliminary work in confocal microscopy has shown that it is possible to simplify diagnosis by using microscopic, in vivo, non-invasive imaging. However, CIM cameras are rare, very expensive and difficult to access.

Conversely, digital dermatoscopes with 400x magnification are much less expensive and can also allow, in a certain number of cases, an examination at the cellular level of tumors, with, in our opinion, the advantage of being easy to learn. In the context of the pooling of resources within medical centers in particular, their dissemination should accelerate. Furthermore, x400 dermatoscopy can provide similar information to IVCM for the most frequent black genital tumors.

DETAILED DESCRIPTION:
The hypothesis that motivates this work is that X400 dermatoscopy in the hands of non-experts would allow a fast increase in their diagnostic capacity by identifying the main genital pigmented tumor, namely melanosis, and thus improve the use of expert centers relieved of the care of benign tumors.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with a pigmented lesion of the genital mucosa, having benefited from a mucosal consultation at the University Hospital of Saint-Etienne, with Professor Perrot.
* The patient's clinical file must contain clinical images, dermatoscopy images x 20 and at least 1 dermatoscopy image x 400.

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women with a pigmented lesion of the genital mucosa will be included.
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Comparison results between expert dermatologists with x20 dermatoscopic photos (Group A) and non-dermatologists physicians with x400 dermatoscopic photos (Group B) | Year: 1
  Performance of x400 dermatoscopic (results of expert dermatologists versus non-dermatologists physicians)

SECONDARY OUTCOMES:
Comparison results between expert dermatologists with x20 dermatoscopic photos (Group A) and gynecologists with x400 dermatoscopic photos (Group B1) | Year: 1
  Performance of x400 dermatoscopic (results of expert dermatologists versus gynecologists)
Comparison results between expert dermatologists with x20 dermatoscopic photos (Group A) and general practitioners with x400 dermatoscopic photos (Group B2) | Year: 1
  Performance of x400 dermatoscopic (results of expert dermatologists versus general practitioners)
Comparison results between gynecologists with x400 dermatoscopic photos (Group B1) and general practitioners with x400 dermatoscopic photos (Group B2). | Year: 1
  Performance of x400 dermatoscopic (results of gynecologists versus general practitioners)
Comparison results between expert dermatologists with x400 dermatoscopic photos (Group A) and skin Artificial intelligence software with x400 dermatoscopic photos (Group C). | Year: 1
  Performance of x400 dermatoscopic (results of expert dermatologists versus skin Artificial intelligence software)
Comparison results between dermatologists physicians with x400 dermatoscopic photos (Group B) and skin Artificial intelligence software with x400 dermatoscopic photos (Group C). | Year: 1
  Performance of x400 dermatoscopic (results of dermatologists physicians versus skin Artificial intelligence software)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Luc Perrot, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No